CLINICAL TRIAL: NCT03057886
Title: COMPARATIVE STUDY BETWEEN THE USE OF THE "SPOT ON" THERMOMETER AND THE ORAL AND ESOPHAGEAL THERMOMETERS IN SPINAL AND GENERAL ANESTHESIA
Brief Title: Study to Evaluate the Accuracy of the New Monitor of Temperature in Comparison With the Consecrated Thermometers by Literature
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ricardo Caio Gracco De Bernardis (Other)
Collaborators: HOSPITAL GERAL DE ITAPECERICA DA SERRA (Unknown)
Responsible Party: Sponsor-Investigator, Ricardo Caio Gracco De Bernardis, PHD, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Organization: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Other Study IDs: 56202616.9.0000.0083
Record Dates: First submitted 2017-02-02; First posted 2017-02-20 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Compare the Spot On with others consecrated thermometers: This study intends to compare the accuracy of the new device(SPOT ON thermometer) with the oral and esophageal in participants submitted to general and spinal anesthesia, in different types of population (pediatric and adult)
  Interventions: Device: Comparative thermometers to compare with a new device

INTERVENTIONS:
Device: Comparative thermometers to compare with a new device — The made up for the choice of the thermometer to be to general anesthesia the oral and new device (Spot On thermometers) before anesthesia induction, after anesthesia induction the Spot On, and oral, and esophageal thermometers and after surgery in PACU the Spot On and oral thermometer. In group submitted to spinal anesthesia the made up for the choice of the thermometer to be the oral and Spot On thermometers before anesthesia induction, after anesthesia induction the Spot On and oral thermometers and after surgery in PACU the Spot On and oral thermometer.

SUMMARY:
This study compares the use of the "SPOT ON" thermometer with the oral, esophageal in participants submitted to general and the oral thermometer to spinal anesthesia, from the pre op, intra and post op stages, evaluating the accuracy of this new monitor against the already consecrated one by literature. The Investigators will analyze in three different types of anesthesia (general, spinal and pediatric population).

DETAILED DESCRIPTION:
After approval by the Institutional Research Ethics Committee, the adults and pediatrics participants for elective surgeries to be submitted to general and spinal anesthesia lasting 60 minutes or more held at the surgery center at Itapecerica of Serra Hospital. The participants will receive the necessary explanations on the research and, after obtaining the responsible consent for participating in the trial, the participants will be included.

Inclusion/exclusion criteria:

Inclusion - adults and pediatrics population that will be submitted to general or spinal anesthesia in the surgery center at Itapecerica of Serra Hospital.

Exclusion:

* The participants that are feverish/present with infectious symptoms
* Refusal of the use of the device by the participants There will be select each groups made up of 70 participants. It will be submitted the adults in two groups, one submitted to general anesthesia and other group submitted to spinal anesthesia and the pediatric group to general anesthesia. The made up for the choice of the thermometer to be to general anesthesia the oral and Spot On thermometers before anesthesia induction, after anesthesia induction the Spot On, and oral, and esophageal thermometers and after surgery in PACU the Spot On and oral thermometer. In group submitted to spinal anesthesia the made up for the choice of the thermometer to be the oral and Spot On thermometers before anesthesia induction, after anesthesia induction and after surgery in PACU the Spot On and oral thermometer.

The thermometer will be used as the moment they will be identified as:

Adult General Group (AGG): the anesthetic procedure will use the spot on thermometer during the pre, intra and post-operative stages and in association with oral during the pre, intra and post-operative stages and the esophagus thermometer during the intra-operative stage.

Adult Spinal Group (ASG): the anesthetic procedure will use the oral and the spot on thermometer in the pre, intra and post-operative stages.

Pediatric General Group (ASG): the anesthetic procedure will use the oral in the pre, intra and post-operative stages and esophageal thermometers in the intra stages and the spot on thermometer during the pre, intra and post-operative stages.

The anesthetic technique will be standard according to the scheduled surgery. The study will assess the participants submitted to elective anesthesia throughout the pre, intra and post-operative stages of all scheduled elective surgeries.

All the participants for elective surgeries lasting 60 minutes or more and/or are scheduled to use any active heating device from the pre, intra and post-anesthetic stages up till the discharge from the post anesthesia recovery room.

The variables to be assessed in the study are:

* Age, gender, weight, height, physical condition according to the American Anesthesiology Association classification;
* Oral, SPOT ON, and esophagus temperature measured at the following points:

  * Mentrance - entering the room and every 10 min until the anesthesia induction
  * Minduction - immediately before induction
  * M10, M20, M30 = 10, 20, 30 min after induction and every 10 min till the end of the anesthetic procedure;
  * Mpost-0, Mpost-15, Mpost-30, Mdischarge, = 0, 15, 30, and every 15 min till the discharge from post anesthesia recovery room.
* Room temperature of operating room and post anesthesia recovery room (from the participants entrance every 30 minutes to the end of the procedure and discharge to the hospital bed).

Data analysis The data will be tabulated and noted as mean and standard deviation, whenever possible, and observed for normal distribution using the Kolmogorov-Smirnov test (sample size exceeding 50). Nonparametric data will be presented by Mid and distribution boundaries. The values of temperatures are compared by estimation model of generalized equations (GEE) with Bonferroni correction (REF: Guimarães and Hirakata, 2012).

The calculation of the sample consider the participants as his own control (intragroup) and also the comparison between the equipment used (between groups, all three). Using multivariate analysis of variance (ANOVA) repeated measures, with test significance level (alpha) 1% (probability of error type I) and sample size which reduces the probability of type II error (Beta) in 95%, the sample is situated on 120 participants(Ref: Faul et al 2007).

ELIGIBILITY:
The participants for elective surgeries to be submitted to general and spinal anesthesia lasting 60 minutes or more held at the central operating center at the Itapecerica da Serra Hospital.

The participants will receive the necessary explanations on the research and, after obtaining the responsible consent for participating in the trial, they will be included.

Inclusion Criteria: adults and pediatrics population that will be submitted to general or spinal anesthesia in the surgery center at Itapecerica of Serra Hospital.

Exclusion Criteria:• Patients that are feverish/present with infectious symptoms and Refusal of the use of the device by the patient

-

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will analyze in three different types of anesthesia and population (general and spinal anesthesia and pediatric and adult population)
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Compare the Spot On temperature and the consecrated termometer in the perioperative term. | 30 weeks
  measure the temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Geral de Itapecerica da Serra, Itapecerica da Serra, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We will publish the data and result after the conclusion of study.

REFERENCES:
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Akata T, Setoguchi H, Shirozu K, Yoshino J. Reliability of temperatures measured at standard monitoring sites as an index of brain temperature during deep hypothermic cardiopulmonary bypass conducted for thoracic aortic reconstruction. J Thorac Cardiovasc Surg. 2007 Jun;133(6):1559-65. doi: 10.1016/j.jtcvs.2006.11.031. PMID 17532957
- [Result] Kimberger O, Thell R, Schuh M, Koch J, Sessler DI, Kurz A. Accuracy and precision of a novel non-invasive core thermometer. Br J Anaesth. 2009 Aug;103(2):226-31. doi: 10.1093/bja/aep134. Epub 2009 May 29. PMID 19482858
- Available data/document: Study Protocol: 56202616.9.0000.0083 — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — There you may find the project and all step to get the approval